CLINICAL TRIAL: NCT05856955
Title: Mobile Health for Enhanced Hypertension Self-Management
Brief Title: Mobile Health Management of Hypertension
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB23-1612; 5K23HL165110-03 (NIH)
Record Dates: First submitted 2023-05-03; First posted 2023-05-12 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enhanced Usual Care (Active Comparator): The active comparison group will receive a smartphone with the WebMD® health information application preloaded and a BP monitor. After recruitment, participants will receive a confirmatory interview, informed consent, and baseline device training via telephone, delivered by an experienced research assistant. Participants will be encouraged to complete 1 morning BP reading daily, irrespective of study arm. BP readings are automatically uploaded via Bluetooth to a centralized, secure platform to be accessible to the study PI.
  Interventions: Behavioral: Enhanced Usual Care
- Behavioral mHealth Coaching Intervention (Experimental): Those randomized to the intervention group will receive a smartphone with the intervention program preloaded in addition to a BP monitor. After recruitment, participants will receive a confirmatory interview, informed consent, and baseline device training via telephone, delivered by an experienced research assistant. Participants will be encouraged to complete 1 morning BP reading daily, irrespective of study arm, however, only the intervention group will receive reminders from the mHealth coaching intervention to check BP daily. BP readings are automatically uploaded via Bluetooth to a centralized, secure platform to be accessible to the study PI.
  Interventions: Behavioral: mHealth Coaching Intervention

INTERVENTIONS:
Behavioral: mHealth Coaching Intervention — The intervention uses a mHealth virtual tool that facilitates human-device interaction and is delivered by smartphone application. The program has coaching and education components that lead to chronic disease behavior change. It has been previously validated to improve self-management, medication adherence, and quality of life in individuals with CVD. The participant engages by selecting responses on the touch screen. In this manner, participants converse with the coach, develop a therapeutic alliance, and record responses. The investigators will institute behavior change methodology to enhance intervention efficacy.
  Arms: Behavioral mHealth Coaching Intervention
Behavioral: Enhanced Usual Care — Smart phone without health coach. A basic health application is installed on the smart phone provided to the participant.
  Arms: Enhanced Usual Care

SUMMARY:
The investigators will pilot test a hypertension self-management intervention for feasibility and acceptability. The investigators will enroll adults (age ≥18) with uncontrolled hypertension, identified from the electronic health record. In this feasibility trial, the research aim is to explore trial design, participant acceptability of the intervention and outcome measures, and to generate data to inform the design of a future randomized controlled trial.

DETAILED DESCRIPTION:
The investigators will pilot test a hypertension self-management intervention for feasibility and acceptability. This is a pilot study to gain experience in enrolling and retaining patients from the identified population and collecting outcome variables. Study cohort: The investigators will enroll adults (age ≥18) with uncontrolled hypertension, identified from the electronic health record problem list and an average systolic blood pressure (BP) of 150-199 or diastolic of 95-119 mmHg at 2 ambulatory visits, 1 of which is within 6 months of study entry. These BP criteria ensure enrollment of individuals who warrant improved BP control. In this feasibility trial, the research aim is to explore trial design, participant acceptability of the intervention and outcome measures, and to generate data to inform the design of a future RCT. We will employ a validated approach to determine feasibility (e.g., acceptability, satisfaction, and practicality).

All secondary measures will be collected at baseline, 30 days, and end of intervention (90 days). These outcomes are pilot measures that will be used in a subsequent full-scale efficacy trial of the intervention.

Study protocol. Duration = 90 days. Allocation will use a randomly permuted block design. The investigators will provide smartphones and cellular subscriptions to all participants, as in their prior studies of cardiovascular disease mobile health interventions. This obviates the need for smartphone ownership or internet access. Participants randomized to the intervention group will receive the smartphone with the intervention program preloaded in addition to a BP monitor. The active comparison group will receive a smartphone with a basic health information application preloaded and a BP monitor. After recruitment, participants will receive a confirmatory interview, informed consent, and baseline device training via telephone, delivered by an experienced research assistant. Participants will be encouraged to complete 1 morning BP reading daily, irrespective of study arm, however, only the intervention group will receive reminders from the mHealth coaching intervention to check BP daily. BP readings are automatically uploaded via Bluetooth to a centralized, secure platform to be accessible to the study PI. Participants will receive $20 for the baseline telephone visit and $40 at study completion. As in the groups' prior RCTs, the final payment requires return of the smartphone.

Sample Size Justification and Recruitment. Investigators will focus on feasibility outcomes among 40 patients, following examples in the literature and guidelines for feasibility studies, which recommend against estimating preliminary efficacy or standard errors using pilot data. Nevertheless, with 40 participants, the investigators will have the ability to calculate point estimates and 95% confidence intervals with a margin of error of 0.22. The cohort of 40 will be reasonably recruited in the allotted timeframe. Culturally sensitive recruitment strategies will be employed to ensure participant diversity. In addition, participants will be recruited from outpatient clinics via HIPAA-compliant, IRB approved protocols. The investigators will deploy IRB-approved virtual recruitment strategies previously developed by the study's PI with study brochure and opt-out postcard; electronic health record screening for eligibility; telephone-based confirmatory interview, and informed consent.

Statistical Analysis. Descriptive data, such as means, standard deviations, and sample proportions, will be reported for all participants and by study arm. Data with non-normal distributions will be transformed, as needed. The primary focus will be on feasibility and acceptability as defined above. Primary outcomes will be assessed with point estimates and 95% CIs. Any between-arm differences will be examined using χ2 tests or 2-sided Fisher's exact test for categorical variables, and 2-tailed t tests for continuous variables. Continuous secondary outcomes (locus of control, resilience, BP) will be analyzed using ANCOVA comparing 90-day outcomes between arms after adjusting for baseline BP. The proportion of participants who are normotensive will be analyzed by logistic regression as a function of study arm.

ELIGIBILITY:
Inclusion Criteria:

* Prescribed use of 1 or more antihypertensive medications
* English-speaking
* Residence in a disadvantaged neighborhood

Exclusion Criteria:

* History of malignant HTN
* Inability to comprehend the study protocol
* Institutionalized status
* Significant sensory or neurocognitive deficit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2027-09 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Participant acceptance and adherence to program | 90 days
  80% of participants receiving intervention will have strong engagement, defined by >60 logins
Participant satisfaction and usability | 90 days post index discharge
  80% of participants receiving intervention will indicate talking with the coach was easy on a 7-point Likert scale (1=Easy; 7=Difficult)
Practicality of participant self-monitoring behavior | 90 days
  80% of participants receiving intervention will have recorded their BP >60 times

SECONDARY OUTCOMES:
Locus of control | 90 days
  a measure of beliefs that one's health is determined by factors either intrinsic or extrinsic to one's self. Uses the 24-item Multidimensional Health Locus of Control.
Resilience | 90 days
  Resilience is an important measure given our asset-based approach signifying that some communities have good health outcomes despite having high predicted risk. Uses Connor-Davidson 10 item Scale wherein higher scores are better. Each item is scored on a 5-point Likert scale from 0 ("not true at all") to 4 ("true nearly all of the time"), and the total score is calculated by summing up all 10 items, resulting in a possible range from 0 to 40, where higher scores indicate greater resilience.
Medication Adherence | 90 days
  3-item self-report adherence measure. Uses Voil's adherence scale wherein higher scores are better.
Blood pressure change | 90 days
  Change in BP results from baseline to day 90. Measured in mmHg.
Blood pressure control | 90 days
  Proportion of participants with normal BP (i.e., <135/<85 mmHg) at day 90

CONTACTS AND LOCATIONS:
Overall Officials: Amber Johnson, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
This award does not meet sponsor criteria for a Data Sharing Plan as the direct costs are <$500,000/year.